CLINICAL TRIAL: NCT03056404
Title: Research for Specific Proteins of Interest for the Serological Diagnosis of Bird Fancier's Lung
Acronym: HYPERSENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: API/2015/66
Record Dates: First submitted 2016-08-10; First posted 2017-02-17 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Avian Hypersensitivity Pneumonitis
MeSH Terms: conditions — Bird Fancier's Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- control subject (Experimental): additional blood sample and 15 control subjects will be seen in consultations in the service of pneumology. The visit will include an auscultation, a respiratory functional exploration and a blood test (2 tubes of 7 ml of total blood). A questionnaire of exhibition will be realized to collect the species of birds and the times of exhibition.
  Interventions: Other: additional blood sample; Other: respiratory functional exploration

INTERVENTIONS:
Other: additional blood sample
Other: respiratory functional exploration

SUMMARY:
This study aims at identifying bird proteins useful for diagnostic tests to determine the cause of Bird Fancier's Lung (BFL).

DETAILED DESCRIPTION:
Allergic diseases are an important part of health concerns in Europe and in countries "industrialized". Among them are distinguished from hypersensitivity pneumonitis (HP), consecutive to repeated inhalation of organic substances (bacteria, fungi, avian proteins ...).

As with other HP, the BFL is a invalidating disease, but usually not lethal if the patient reduced sufficiently early exposure to antigens.

Associated symptoms include breathing difficulties a dry cough, a general fatigued state accompanied by a fever and a rapid and pronounced weight loss.

These clinical signs may be similar to a flu-like condition, difficult to discern from other respiratory disease. Diagnosis is based on a set of clinical, radiological and biological arguments that are often discussed.

Using these criteria as predictors would increase opportunities to diagnose HP without using invasive clinical examinations such as biopsy and bronchoalveolar lavage.

Although serology is a useful argument for the diagnosis, its value is often criticized.

Thus, significant variations in performance of serological tests are observed from one provider to another and, for the same supplier, from one batch to another.

This issue could be raised by the use of recombinant antigens. The principle is to use only to the reaction the purified protein of interest produced by genetic engineering.

The Parasitology-Mycology department has acquired expertise in the research of proteins of interest for serology allergic diseases and in the manufacture of recombinant antigens. Thus the work of the team have identified proteins of interest for the diagnosis of two HP of occupational origin and translates this expertise to identify pigeon's proteins and study the feasibility of this research.

For this project, the pigeon droppings (Columba livia), collected from different breeders in the region were identified as antigenic source.

The objective of the HYPERSENS project is to extend the problematic to other species of birds and understand the specific species of antigenic proteins. The aim is also to identify and produce recombinant proteins that will identify the cause of avian hypersensitivity pneumonitis.

ELIGIBILITY:
Inclusion criteria:

* Exposure known about birds
* Non-smoker
* Absence of compatible respiratory symptoms with a HP

Exclusion Criteria:

* Farmer,
* smoker,
* pregnancy and feeding,
* minor subject,
* known immunizing deficit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
number of protein of interest | 24 months
  5 and 15 proteins for all selected birds

SECONDARY OUTCOMES:
Selection and identification of protein of interest specific for each selected bird | 24 months
  Identifying at least three specific proteins for each bird species by 2D-Electrophoresis and Western blotting (based on previous study).
Selection and identification of proteins of interest common to all selected bird'droppings | 24 months
  Identifying at least one common protein to all droppings of selected bird species by 2D-Electrophoresis and Western blotting. This protein will be recognized by the antibodies of all patients regardless of their exposure and not recognized by controls. It would make the diagnosis of BFL for any avian exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Millon, Principal Investigator — lmillon@chu-besancon.fr
Locations (1):
- Centre Hospitalier Régional Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rouzet A, Reboux G, Dalphin JC, Gondouin A, De Vuyst P, Balliau T, Millon L, Valot B, Roussel S. An immunoproteomic approach revealed antigenic proteins enhancing serodiagnosis performance of bird fancier's lung. J Immunol Methods. 2017 Nov;450:58-65. doi: 10.1016/j.jim.2017.07.012. Epub 2017 Jul 29. PMID 28760669